CLINICAL TRIAL: NCT00164840
Title: Symptomatic Gastroesophageal Reflux Disease: Double Blind Randomized Controlled Study of On-demand Therapy Versus Maintenance Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OG Study
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2010-03-30 (Estimated); Status verified 2010-03

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: GERD
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Esomeprazole

INTERVENTIONS:
Drug: Esomeprazole

SUMMARY:
Maintenance treatment with proton pump inhibitor (PPI) is the most widely recommended modality of treatment for long-term management of gastroesophageal reflux disease (GERD). Yet in clinical practice treatment is commonly given in short courses on as required basis during symptom flare up, particularly for patients with mild to moderate GERD.

On-demand therapy also has the potential advantage that patient does not need to take regular medications, thereby improving the quality of life. However, whether on-demand PPI therapy achieves similar efficacy of symptom control is uncertain.

The aim of this study is to compare the efficacy and quality of life of on-demand and maintenance PPI regimens in long-term management of non-erosive GERD patients. The investigators hypothesize that on-demand PPI treatment is as effective as maintenance PPI.

ELIGIBILITY:
Inclusion Criteria:

* Weekly symptoms of heartburn or acid regurgitation of moderate severity as predominant complaint for at least 6 months

Exclusion Criteria:

* Erosive esophagitis
* Concomitant peptic ulcer disease
* Use of NSAID in recent 4 weeks (Low dose aspirin < 300 mg is allowed)
* Pregnant or lactating female
* Illiterate patient (who cannot administer questionnaire)
* Known hypersensitivity to PPI

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2003-05; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Treatment failure | 26 Weeks

SECONDARY OUTCOMES:
Symptom score | 26 weeks
Quality of Life | 1 year
Number of days off treatment

CONTACTS AND LOCATIONS:
Overall Officials: Justin CY WU, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Endoscopy Centre, Prince of Wales Hospital, Hong Kong, China